CLINICAL TRIAL: NCT04330950
Title: A Preliminary Study of the Incidence, Risk Factors and Sequelae of Postoperative Delirium in Elderly Patients Undergoing Major Non-Cardiac Surgery in Singapore
Brief Title: Postoperative Delirium in Elderly Patients Undergoing Major Non-Cardiac Surgery in Singapore
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/00703
Record Dates: First submitted 2020-03-27; First posted 2020-04-02 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Delirium
Keywords: Geriatrics; Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Cohort: Preoperative: Battery of neurocognitive tests and questionnaires (MoCA, PHQ-9, Falls History, FIFE, STOPBANG, Nutritional Survey) Postoperative in PACU: NuDESC test Postoperative 30 days: 10 minute phone interview
  Interventions: Other: Neurocognitive tests

INTERVENTIONS:
Other: Neurocognitive tests — Preoperative: Battery of neurocognitive tests and questionnaires (MoCA, PHQ-9, Falls History, FIFE, STOPBANG, Nutritional Survey) Postoperative in PACU: NuDESC test Postoperative 30 days: 10 minute phone interview

SUMMARY:
The primary aim of this study is to investigate the incidence, risk factors and sequelae of postoperative delirium in elderly patients undergoing major non-cardiac surgery in Singapore. The secondary aim of this study is to look for EEG markers of POD that may potentially lead to the development of a POD monitor.

DETAILED DESCRIPTION:
Singapore's population is growing older and increasingly burdened with systemic disease. It is estimated that over 320 million people underwent surgery worldwide in 2010, with Asia being the fastest growing region. Elderly patients aged >65 years are presenting for surgery at an ever-increasing rate. In the United States, studies have estimated that approximately 53% of all surgical procedures are performed on patients over the age of 65. Projections estimate that approximately half of the population over the age of 65 will require surgery once in their lives.

It is recognized that for elderly patients, quality of life after surgery matter more than quantity of life. Elderly patients have diminished reserves and poorer recovery potential. Therefore, to fully benefit from surgery, it is essential to adopt measures to preserve quality of life in addition to survival after surgery in the perioperative period. One example is the enhanced recovery after surgery (ERAS) programme where protocolized care involving optimal analgesia, less invasive surgeries, early mobilisation and early hospital discharge has improved the recovery of patients after surgery. In the best practice guidelines for care of elderly surgical patients put forward by the American College of Surgeons National Surgical Quality Improvement Program (ACS NSQIP) and the American Geriatrics Society (AGS) published in 2012, anaesthesia plays a role in more than half of the 13 recommendations put forward.

One of these recommendations is to reduce postoperative delirium (POD). The anaesthetic agents we use is toxic to the brain, and deep anaesthesia causes POD, which is linked to increased hospital length of stay, unplanned hospital readmissions, increased 30-day mortality, and dementia. POD is one of the leading causes of why patients fall at home after surgery. Up to 10% will develop long-term neurocognitive deficits, which in turn diminish the quality of life and levy a tremendous socio-economic burden on family and care-givers, and shortens life. The topic of POD has dominated the anaesthesia literature in the last year, with both the US and European societies issuing best practice guidelines such as the Brain Health Initiative and the Safe Brain Initiative, as well as harmonization of the definitions of postoperative neurological outcomes with that used by neurologists in compliance with DSM-5 definitions to allow for collaborative solutions.

More recently it was reported in the Straits Times that Singaporeans have the longest life expectancy in the world. However, 10.7 years of this is spent in poor health, with diminished mental health ranking as the second most important cause for this. Because POD is strongly linked to the development of dementia and/or alters the trajectory at which age-related dementia occurs, it is very important to prevent the development of POD. This is particularly so as studies have shown that POD is very common, occurring in as many as 11-50% of patients undergoing major non-cardiac surgery, and that up to 40% of POD is preventable.

Awareness of POD remains poor amongst both doctors and the public. The reason for this is that POD requires specialized neurological testing and currently, there are no established biomarkers or monitors to detect it. Anecdotally, POD is one of the leading reasons for in-hospital (blue letter) psychiatric referrals after surgery in NUHS, as delirious patients will refuse to comply with physiotherapy, medications and wound care, leading to delayed healing, infection and delayed discharge. Patients are not routinely assessed for POD and can be discharged from hospital with it. Patients who are still delirious can end up with poor feeding and self-care, and even hurt themselves leading to rehospitalisation. In short, POD is a common yet under-diagnosed, and potentially preventable, complication of anaesthesia and surgery in the elderly that has significant long-term effects on the independence of patients after surgery and their quality of life.

The current accepted standard for diagnosing POD is to perform twice daily neurocognitive assessments daily in the first 5 postoperative days. However, as this is difficult to implement due to the significant manpower requirements, delirium in the post-anaesthesia care unit (PACU delirium) has been used as a surrogate for POD. PACU delirium is distinct from emergence delirium which occurs upon arrival or soon after admission into the PACU and is related to residual effects of anaesthesia. Emergence delirium typically is self-limiting and has no long-term sequelae. In contrast, PACU delirium occurs after recovery from the effects of anaesthesia, presenting at 30-60 minutes after arrival in the PACU. PACU delirium occurs in up to 80% of patients who subsequently develop POD in the wards and has been independently associated with increased length of hospitalization, unplanned readmission, and increased in-hospital mortality.

Therefore, the primary aim of this study is to investigate the incidence, risk factors and sequelae of postoperative delirium in elderly patients undergoing major non-cardiac surgery in Singapore. The secondary aim of this study is to look for EEG markers of POD that may potentially lead to the development of a POD monitor. This study will provide preliminary data to enable the investigators to apply for a national grant for a more definitive and adequately powered study. It is envisaged that eventually, the information gathered will allow the investigators to form an effective clinical plan to reduce postoperative delirium in our elderly patients undergoing non-cardiac surgery, and a basis to apply for national grant funding to implement the clinical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients aged 65 and above
* Undergoing major non-cardiac surgery, defined as a surgery that is at least 2 hours in duration and requiring at least 1 day postoperative stay in hospital

Exclusion Criteria:

* Undergoing emergency surgery
* Undergoing surgery under local anaesthesia
* History of psychiatric disease
* Illiterate
* Active history of substance abuse
* Undergoing neurosurgical procedures
* A second surgery planned within 5 days of index surgery
* Non-resident of Singapore
* Deaf, dumb or mute
* Patients planned for admission into the Intensive Care Unit after surgery
* Pregnant women

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients aged 65 and above who are planned for major non-cardiac surgery of at least 2 hours in duration and requiring at least 1 postoperative stay in hospital.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Investigate the incidence, risk factors and sequelae of postoperative delirium in elderly patients undergoing major non-cardiac surgery in Singapore | After surgery through to postoperative day 30
  By collecting the patient's demographics, medical records and surgical records, and looking at their outcome, we aim to investigate the incidence and risk factors of postoperative delirium in this elderly cohort in Singapore

SECONDARY OUTCOMES:
Look for EEG markers of POD that may potentially lead to the development of a POD monitor | Postoperative through study completion, an average of 1 year
  Look for EEG markers of POD that may potentially lead to the development of a POD monitor

CONTACTS AND LOCATIONS:
Overall Officials: Lian Kah Ti, Principal Investigator — National University Health System
Locations (4):
- Singapore (4):
  - Khoo Teck Puat Hospital, Singapore
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rose J, Weiser TG, Hider P, Wilson L, Gruen RL, Bickler SW. Estimated need for surgery worldwide based on prevalence of diseases: a modelling strategy for the WHO Global Health Estimate. Lancet Glob Health. 2015 Apr 27;3 Suppl 2(Suppl 2):S13-20. doi: 10.1016/S2214-109X(15)70087-2. PMID 25926315
- [Background] Yang R, Wolfson M, Lewis MC. Unique Aspects of the Elderly Surgical Population: An Anesthesiologist's Perspective. Geriatr Orthop Surg Rehabil. 2011 Mar;2(2):56-64. doi: 10.1177/2151458510394606. PMID 23569671
- [Background] Aldecoa C, Bettelli G, Bilotta F, Sanders RD, Audisio R, Borozdina A, Cherubini A, Jones C, Kehlet H, MacLullich A, Radtke F, Riese F, Slooter AJ, Veyckemans F, Kramer S, Neuner B, Weiss B, Spies CD. European Society of Anaesthesiology evidence-based and consensus-based guideline on postoperative delirium. Eur J Anaesthesiol. 2017 Apr;34(4):192-214. doi: 10.1097/EJA.0000000000000594. PMID 28187050
- [Background] Evered L, Silbert B, Knopman DS, Scott DA, DeKosky ST, Rasmussen LS, Oh ES, Crosby G, Berger M, Eckenhoff RG; Nomenclature Consensus Working Group. Recommendations for the nomenclature of cognitive change associated with anaesthesia and surgery-2018. Br J Anaesth. 2018 Nov;121(5):1005-1012. doi: 10.1016/j.bja.2017.11.087. Epub 2018 Jun 15. PMID 30336844
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] American Geriatrics Society Expert Panel on Postoperative Delirium in Older Adults. Postoperative delirium in older adults: best practice statement from the American Geriatrics Society. J Am Coll Surg. 2015 Feb;220(2):136-48.e1. doi: 10.1016/j.jamcollsurg.2014.10.019. Epub 2014 Nov 14. No abstract available. PMID 25535170